CLINICAL TRIAL: NCT06340958
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Parallel-Design, Phase 2 Study to Assess the Efficacy and Safety of CLE-100 as an Adjunctive Treatment for Major Depressive Disorder Patients With Inadequate Response to Standard Antidepressants
Brief Title: A Study of CLE-100 (Oral Esketamine) as an Adjunctive Treatment to Standard Antidepressants for Major Depressive Disorder
Acronym: SOLEO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Clexio Biosciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLE100-MDD-202
Record Dates: First submitted 2024-03-25; First posted 2024-04-02 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Adjunctive Treatment of Major Depressive Disorder (MDD)
Keywords: MDD, inadequate response, depression, depressive disorder, major depression, adjunct therapy, oral, esketamine
MeSH Terms: conditions — Depression; Depressive Disorder; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CLE-100 (Experimental): 1 oral tablet of CLE-100 once daily (in addition to current anti-depressant drug) for 4 weeks
  Interventions: Drug: CLE-100
- Placebo (Placebo Comparator): 1 oral tablet of Placebo once daily (in addition to current anti-depressant drug) for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CLE-100 — 1 tablet of CLE-100 administered once daily
  Arms: CLE-100
Drug: Placebo — 1 tablet of placebo administered once daily
  Arms: Placebo

SUMMARY:
The study is a Phase 2, double-blind, randomized, placebo-controlled study in Major Depressive Disorder (MDD) participants with an inadequate response to standard antidepressants The objective of the study is to assess CLE-100 (oral esketamine) for the treatment of MDD in participants currently treated with an oral antidepressant medication and who have an inadequate response to at least 2 antidepressants.

DETAILED DESCRIPTION:
This is a Phase 2 study in subjects with MDD currently treated with an oral antidepressant medication with an inadequate response to at least 2 antidepressants. SOLEO will be an outpatient study to assess the safety, efficacy, and tolerability of CLE-100 as compared to placebo.

Eligible subjects will be randomized to receive either placebo or CLE-100 (oral esketamine) once daily in addition to their current oral antidepressant monotherapy for 4 weeks. All subjects who adequately completed the 4-week Double-Blind Treatment Period and who meet the eligibility criteria will be offered the option to roll-over to a 6-month Open-label Extension (OLE) Treatment Period with CLE-100.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 to 65 years of age at Screening
2. Diagnosis of MDD, single or recurrent, without psychotic features, in the current or previous episode(s), according to the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5). The diagnosis of MDD must be supported by the Mini International Neuropsychiatric Interview (MINI) Screen 7.0.2 for DSM-5.
3. Currently experiencing a Major Depressive Episode (MDE) that began at least 12 weeks but no more than 5 years prior to Screening. The current MDE must be confirmed by the independent SAFER assessor.
4. MADRS score of 24 or higher at Screening as confirmed by an independent SAFER assessor.
5. At Screening, a history of inadequate response to at least 2 antidepressant medications in the current MDE. Inadequate response is defined as less than 50% improvement of depression symptoms following at least 6 weeks of treatment with a therapeutic dose and is assessed by the site using the Massachusetts General Hospital Antidepressant Treatment Response Questionnaire (MGH-ATRQ). Inadequate response to at least 2 antidepressant medications must be verified by documented medical or pharmacy records and confirmed by an independent SAFER assessor.
6. Able and competent to read and sign the informed consent form (ICF).

Exclusion Criteria:

1. At Screening, a history of inadequate response (as defined in inclusion criterion #5) to more than 5 antidepressant medications in the current MDE using MGH-ATRQ and confirmed by the independent SAFER assessor.
2. A high risk of suicide based on any of the following:

   1. Item 10 of MADRS score (suicidal thoughts) is 5 or higher at Screening or Baseline.
   2. Suicide attempt in the previous 6 months.
   3. Significant risk, as judged by the Investigator, based on the psychiatric interview or information collected with the C SSRS at Screening or Baseline.
3. Current or lifetime history of substance use disorder with ketamine, phencyclidine (PCP), lysergic acid diethylamide (LSD), or 3.4-methylenedioxymethamphetamine (MDMA) hallucinogen-related use disorders or has any other current substance use disorder or history within 12 months prior to Screening (Substance Use Disorder is diagnosed per DSM-5 criteria and does not include tobacco use disorder).
4. Use of ketamine, esketamine, PCP, or dextromethorphan recreationally in the past 6 months.
5. History or current diagnosis of bipolar disorder, schizophrenia, or schizoaffective disorder or other schizophrenia spectrum disorders.
6. Dementia, delirium, amnesia, or any other significant cognitive disorder.
7. Any medical condition for which an increase in blood pressure or intracranial pressure or intraocular pressure or tachycardia poses a serious risk (e.g., aneurysmal vascular disease, arteriovenous malformation, or history of intracerebral hemorrhage).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) score | 29 days
  The MADRS is a validated clinician-administered measurement of depression severity commonly used in clinical trials of depression treatments to select subjects and assess efficacy. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.

SECONDARY OUTCOMES:
Change from Baseline in the Clinical Global Impression - Severity (CGI-S) | 29 days
  The CGI-S is a well-known and frequently used clinician-administered instrument for the assessment of MDD that weighs the clinical impact of the identified symptom(s) on behavior and function. The CGI-S grades measures of psychopathology on a scale from 1 to 7.
Change from Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) score | 2 weeks
  The MADRS is a validated clinician-administered measurement of depression severity commonly used in clinical trials of depression treatments to select subjects and assess efficacy. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.
Safety Outcomes: Assessment of the safety and tolerability of CLE-100 compared to placebo | Through study completion, an average of 7 months
  Assessment of the safety and tolerability of CLE-100 compared to placebo using the following assessments:
  * Adverse Events (AEs)
  * Adverse events of special interest (AESIs)
  * Clinical laboratory evaluations
  * Vital signs
  * 12-lead electrocardiogram
  * Modified Observer's Assessment of Alertness/Sedation scale (MOAA/S)
  * Clinician-Administered Dissociative State Scale (CADSS)
  * Incidence of suicidal ideation or behavior as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS)
  * 4-item Brief Psychiatric Rating Scale (BPRS)
  * 20-item Physician Withdrawal Checklist (PWC-20)
  * Bladder Pain/Interstitial Cystitis Symptom Score (BPIC-SS)
  * Digit Symbol Substitution Test (DSST)
  * Discontinuation rates and reason(s) for discontinuation

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Clinical Site 139, La Jolla, California
  - Clinical Site 131, Lafayette, California
  - Clinical Site 130, Upland, California
  - Clinical Site 102, Hollywood, Florida
  - Clinical Site 105, Lauderhill, Florida
  - Clinical Site 140, Miami Springs, Florida
  - Clinical Site 132, Pensacola, Florida
  - Clinical Site 118, Atlanta, Georgia
  - Clinical Site 138, Marietta, Georgia
  - Clinical Site 114, Savannah, Georgia
  - Clinical Site 127, Chicago, Illinois
  - Clinical Site 120, Elgin, Illinois
  - Clinical Site 108, Gaithersburg, Maryland
  - Clinical Site 116, Flowood, Mississippi
  - Clinical Site 126, O'Fallon, Missouri
  - Clinical Site 101, Toms River, New Jersey
  - Clinical Site 103, Beachwood, Ohio
  - Clinical Site 119, North Canton, Ohio
  - Clinical Site 135, Oklahoma City, Oklahoma
  - Clinical Site 107, Austin, Texas
  - Clinical Site 137, Plano, Texas
  - Clinical Site 117, Murray, Utah
  - Clinical Site 115, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No